CLINICAL TRIAL: NCT07159893
Title: Study of Inectolizumab Combined With Steroid Hormone Adjustment Strategies in Treatment-naive Patients With Neuromyelitis Optica Spectrum Disease
Brief Title: Inectolizumab With Steroid Optimization in Newly Treated NMOSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-076
Record Dates: First submitted 2025-07-10; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Neuromyelitis Optica; Autoimmune Diseases; Demyelinating Autoimmune Diseases, CNS
MeSH Terms: conditions — Neuromyelitis Optica; Autoimmune Diseases; Demyelinating Autoimmune Diseases, CNS | interventions — inebilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inebilizumab with Rapid Steroid Tapering group (Experimental): Participants receive:
  1. Acute-phase: Methylprednisolone 1.0g IV daily (Days 1-5)
  2. Maintenance-phase:
     * Day 6: Prednisone 60mg po daily + Inebilizumab 300mg IV
     * Day 20: Second inebilizumab 300mg IV + Prednisone reduced to 60mg po every other day
  3. Steroid tapering schedule:Day 34→30mg EOD → Day 48→15mg EOD → Day 62→10mg EOD → Day 76→5mg EOD → Day 90→Discontinue
  4. Long-term: Third inebilizumab 300mg IV at Week 24
  Interventions: Drug: Inebilizumab + Rapid Steroid Tapering group
- Inebilizumab with Standard Steroid Tapering group (Active Comparator): Participants receive:
  1. Acute-phase (Days 1-5):Methylprednisolone 1.0g IV daily
  2. Maintenance-phase:
     * Day 6: Prednisone 60mg po daily +First inebilizumab 300mg IV
     * Day 20: Second inebilizumab 300mg IV+Continue prednisone 60mg po daily until Day 34
  3. Steroid Tapering Schedule:
     Day 34→60mg EOD → Day 62→30mg EOD → Day 90→15mg EOD → Day 118→10mg EOD → Day 146→5mg EOD → Day 174→Discontinue
  4. Long-term: Third inebilizumab 300mg IV at Week 24
  Interventions: Drug: Inebilizumab + Standard Steroid Tapering group

INTERVENTIONS:
Drug: Inebilizumab + Rapid Steroid Tapering group — Drug 1: Inebilizumab Generic Name: Inebilizumab Formulation: Injection (Intravenous) Dose: 300 mg Frequency:Day 6 (Week 0): First dose ；Day 20 (Week 2): Second dose ；Week 24: Third dose Route: Intravenous infusion Drug 2: Prednisone Generic Name: Prednisone Formulation: Tablet (Oral) Dose & Tapering:Day 6-19: 60 mg daily；Day 20: 60 mg every other day (EOD)
  ；Day 34: 30 mg EOD → Day 48: 15 mg EOD → Day 62: 10 mg EOD → Day 76: 5 mg EOD → Day 90: Discontinue Route: Oral
  Other Names: Inebilizumab with rapid glucocorticoid taper group
  Arms: Inebilizumab with Rapid Steroid Tapering group
Drug: Inebilizumab + Standard Steroid Tapering group — Drug 1: Inebilizumab Generic Name: Inebilizumab Formulation: Injection (Intravenous) Dose: 300 mg Frequency:Day 6 (Week 0): First dose ；Day 20 (Week 2): Second dose ；Week 24: Third dose Route: Intravenous infusion Drug 2: Prednisone Generic Name: Prednisone Formulation: Tablet (Oral) Dose & Tapering:Day 6-34: 60 mg daily;Day 34: 60 mg EOD → Day 62: 30 mg EOD → Day 90: 15 mg EOD → Day 118: 10 mg EOD → Day 146: 5 mg EOD → Day 174:Discontinue; Route: Oral
  Other Names: Inebilizumab with standard glucocorticoid taper group
  Arms: Inebilizumab with Standard Steroid Tapering group

SUMMARY:
Title: Study of Inectolizumab Combined With Steroid Hormone Adjustment Strategies in Treatment-naive Patients With Neuromyelitis Optica Spectrum Disease Objective:This study aims to evaluate the steroid-sparing effect and safety of inebilizumab in treatment-naïve AQP4-IgG seropositive neuromyelitis optica spectrum disorder (NMOSD) patients, while assessing its impact on EDSS score improvement during acute-phase treatment. The study will further explore treatment-related biomarkers, including dynamic changes in: immunoglobulin levels, lymphocyte subset profiles, serum AQP4-IgG titers, glial fibrillary acidic protein (GFAP), and neurofilament light chain (NFL) levels.

Study Design:This is a single-center, randomized, open-label, prospective clinical study planning to enroll 25 treatment-naïve, anti-aquaporin-4 immunoglobulin G (AQP4-IgG) seropositive neuromyelitis optica spectrum disorder (NMOSD) patients.

DETAILED DESCRIPTION:
Research Objectives:

* To investigate the steroid-sparing effect and safety of inebilizumab in treatment-naïve AQP4-IgG-positive neuromyelitis optica spectrum disorder (NMOSD) patients.
* To evaluate the efficacy of early inebilizumab initiation during acute attacks in improving EDSS scores and its safety profile in treatment-naïve AQP4-IgG+ NMOSD patients.

Research Background: Neuromyelitis optica spectrum disorder (NMOSD) is a rare, relapsing autoimmune disease characterized by inflammatory demyelination of the central nervous system, predominantly affecting young to middle-aged women and typically manifesting as optic neuritis and longitudinally extensive transverse myelitis, often causing irreversible neurological damage and significant disability. The pathogenesis centers on AQP4-IgG-mediated immune attacks through complement-dependent cytotoxicity and antibody-dependent cell-mediated cytotoxicity, leading to astrocyte damage and neuroinflammation, with B cells and IL-6 playing key roles in disease progression. While traditional therapies (corticosteroids and immunosuppressants) have limited efficacy and significant side effects, newly approved biologics (inebilizumab, eculizumab, satralizumab) targeting B cells, complement, or IL-6 pathways have shown promising results in reducing relapses. Our preliminary data suggest early inebilizumab initiation during acute attacks (within 7-10 days) may improve neurological function (EDSS scores) while enabling rapid steroid tapering without increasing relapse risk. This study aims to systematically evaluate the feasibility and safety of accelerated steroid reduction during inebilizumab therapy in treatment-naïve AQP4-IgG+ NMOSD patients, while assessing the efficacy of early biologic intervention, with the goal of optimizing treatment strategies, improving patient outcomes, and informing future clinical guidelines.

Research Design: This prospective, randomized controlled trial will evaluate the steroid-sparing efficacy and safety profile of inebilizumab in treatment-naïve AQP4-IgG+ neuromyelitis optica spectrum disorder (NMOSD) patients. The study specifically aims to: (1) quantify inebilizumab's glucocorticoid dose-reduction potential, (2) assess its safety in acute-phase administration (initiated within 7-10 days of disease onset), and (3) measure treatment impact on disability outcomes (EDSS improvement). By systematically investigating whether early biologic intervention facilitates both rapid steroid tapering and neurological recovery, this research will generate critical evidence to optimize precision therapy for NMOSD patients.

Treatment Protocol：

Eligible NMOSD patients (n=25) will be randomized into two groups:

* Experimental Group(n=12): Inebilizumab on Day 1 and Day 15. Oral steroids (60 mg qod)after second dose, halved every 2 weeks, stopped at Week 12.
* Active comparator(n=13): Inebilizumab on Day 1 and Day 15. Oral steroids (60 mg qod) after second dose, halved every 4 weeks, stopped at Week 24.

Initial Treatment (Both Groups):

Days 1-5 (D1-D5): Methylprednisolone 1.0g IV daily (first infusion day designated as D1)；Day 6 (D6): Switch to oral prednisone 60mg daily for 14 days + initiate first inebilizumab 300mg IV infusion ；Day 20 (D20): Second inebilizumab 300mg IV (15 days after first dose)；Week 24: Third inebilizumab 300mg IV

Steroid Tapering Schedules:

- Rapid-Taper Group: D20: Prednisone reduced to 60mg every other day (EOD) D34 (after 2 weeks): Reduce to 30mg EOD D48 (after 2 weeks): Reduce to 15mg EOD D62 (after 2 weeks): Reduce to 10mg EOD D76 (after 2 weeks): Reduce to 5mg EOD D90 (Week 12): Discontinue steroids

- Standard-Taper Group: D20-D34: Continue prednisone 60mg daily for 4 weeks D34: Reduce to 60mg EOD D62 (after 4 weeks): Reduce to 30mg EOD D90 (after 4 weeks): Reduce to 15mg EOD D118 (after 4 weeks): Reduce to 10mg EOD D146 (after 4 weeks): Reduce to 5mg EOD D174 (Week 24): Discontinue steroids

Study Visits and Assessments:

* Five scheduled visit timepoints Baseline (Visit 1, Week 0): First inebilizumab administration Visit 2 (Week 2) Visit 3 (Week 4) Visit 4 (Week 12) Visit 5 (Week 24)
* Visit Procedures Visit 1:Laboratory tests (CBC, biochemistry, IgA/IgM/IgG levels, lymphocyte subsets)、MRI (brain/orbital/spinal)、Serum markers (AQP4-IgG, NFL, GFAP)、Clinical assessments (EDSS, Hauser Ambulation Index) Visit 2:Adverse event assessment Laboratory tests (CBC, biochemistry, IgA/IgM/IgG, lymphocyte subsets)、Clinical assessments Visit 3:Adverse event assessment、Clinical assessments Visit 4:Adverse event assessment Laboratory tests (CBC, biochemistry, IgA/IgM/IgG, lymphocyte subsets, serum markers)、Clinical assessments Visit 5:Full repeat of Visit 1 assessments

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the 2015 International Consensus Diagnostic Criteria for Neuromyelitis Optica Spectrum Disorder (NMOSD) and are AQP4-IgG positive, with a first-attack episode;
* Male or female,age >=18 and <=65 years old;
* EDSS score ≤ 7.5;
* Female subjects of childbearing potential must have a negative pregnancy test result during the screening period and must use effective contraception throughout the study period;
* Voluntarily sign the informed consent form.

Exclusion Criteria:

* Laboratory abnormalities include: (white blood cell count < 3×10⁹/L), (neutrophils < 1.5×10⁹/L), (hemoglobin < 85 g/L), (platelet count < 80×10⁹/L), (serum creatinine > 1.5×ULN), (total bilirubin > 1.5×ULN), (AST (GOT) > 3×ULN), (ALT (GPT) > 3×ULN), (alkaline phosphatase > 2×ULN).
* Patients currently suffering from active hepatitis or with a history of severe liver disease are ineligible. Based on the following serological test results for HBsAg, anti-HBc antibodies, and anti-HBs antibodies, there is evidence of hepatitis B virus (HBV) infection: Patients with positive HBsAg should be excluded. For patients with negative HBsAg but positive anti-HBc antibodies, regardless of whether anti-HBs antibodies are positive or negative, HBV-DNA testing is required to determine their status: If HBV-DNA is positive, the patient should be excluded; if HBV-DNA is negative, the patient may be eligible for the trial.
* Patients with other chronic active immune system diseases, or those with stable conditions but requiring glucocorticoid therapy, are excluded, except for neuromyelitis optica spectrum disorder (NMOSD). Examples include rheumatoid arthritis, scleroderma, Sjögren's syndrome, ulcerative colitis, AIDS, genetic immunodeficiency, or drug-induced immunodeficiency. Patients with only positive autoantibodies but without clinical manifestations may be eligible for the trial.
* Pregnant women, breastfeeding women, and patients who plan to conceive during the trial period.
* Allergic reactions: Patients with a history of allergies to contrast agents administered via the parenteral route or to human-derived biological products.
* Patients who received a live vaccine, except for the herpes zoster vaccine, within 28 days prior to randomization.
* Patients who have used rituximab or other monoclonal antibodies within 6 months prior to randomization
* Patients who have received intravenous immunoglobulin (IVIG) within 28 days prior to randomization.
* Patients who have undergone hematopoietic stem cell transplantation or lymphocyte irradiation before randomization.
* Patients who have used immunosuppressive agents such as azathioprine (Azathioprine, AZA, half-life t1/2 = 6 hrs), mycophenolate mofetil (Mycophenolate Mofetil, t1/2 = 16 hrs), leflunomide (Leflunomide, LEF, t1/2 = 14.7 hrs), tacrolimus (Tacrolimus, t1/2 = 43 hrs), teriflunomide (Teriflunomide, t1/2 = 18 days), cyclosporine (Cyclosporin, CsA, t1/2 = 27 hrs), methotrexate (Methotrexate, MTX, t1/2 = 14 hrs), mitoxantrone (Mitoxantrone, NVT, t1/2 = 37 hrs), and cyclophosphamide (Cyclophosphamide, CTX, t1/2 = 6 hrs) before randomization are excluded. Except for leflunomide and teriflunomide, patients can be enrolled if the washout period exceeds five half-lives. For leflunomide and teriflunomide, patients need to undergo cholestyramine washout as follows: take 8 grams of cholestyramine orally three times daily for 11 days. If the 8-gram dose is not tolerated, it can be changed to 4 grams per dose, with the same frequency and duration.
* Patients who have received any investigational drug within 28 days or five half-lives of the trial drug (whichever is shorter) before randomization.
* Patients with symptoms of severe mental illness who are clinically unable to co-operate;
* Patients with malignant tumours.
* Patients who have experienced any of the following events within 12 weeks prior to randomization: myocardial infarction, unstable ischemic heart disease, stroke, or New York Heart Association (NYHA) Class IV heart failure.
* Patients with herpes zoster infection, positive for HCV antibodies, or positive for HIV antibodies during the screening period.
* Patients who are unable to undergo magnetic resonance imaging (MRI) during the trial period.
* Patients whom the investigator deems unsuitable for participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The change in the average daily dose of corticosteroids between the two groups during the follow-up period compared to randomization (i.e., baseline | Baseline, Week 2, Week 4, Week 12, Week 24
  Record the corticosteroid dose for patients at randomization (baseline) and during the follow-up period
Time to first clinical relapse | From the date of randomization (baseline) to the date of first documented clinical relapse (as defined by protocol criteria), assessed up to 24 weeks.
  Accurately document the time of symptom onset in patients.

SECONDARY OUTCOMES:
The change in EDSS (Expanded Disability Status Scale) score from. | Baseline,Week 2, Week 4, Week 12, Week 24
  Before patients enter the study (i.e., at randomization) and at each follow-up time point during the study period, the disability status of patients is assessed by a trained neurologist or study nurse, and the EDSS scores at baseline and follow-up time points are recorded.
The incidence, severity, and outcomes of adverse events in each group of patients | Baseline, Week 2, Week 4, Week 12, Week 24
  Record the occurrence, severity, and outcomes of adverse events in patients at baseline and follow-up time points.
Area Under the Dose-Time Curve of Corticosteroids (AUDTC) | Week 24
  Record the corticosteroid dose for patients at Week 24. Calculate the total area under the dose-time curve (AUDTC) by dividing the dose-time curve into multiple trapezoids, calculating the area of each trapezoid, and then summing these areas.
The change in the Hauser Walking Index from baseline for each group of patients. | Baseline, Week 2, Week 4, Week 12, Week 24
  At baseline and follow-up time points, patients are required to walk 25 feet (approximately 8 meters) on a flat surface, and the time taken is recorded. The score is then determined according to the time taken to walk this distance and whether any assistive devices are used, in accordance with the scoring criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhang, Bachelor, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University

IPD SHARING:
Plan to Share IPD: No